CLINICAL TRIAL: NCT05393167
Title: Pattern of Congenital Anomalies in Infants of Diabetic Mother .
Brief Title: Congenital Anomalies in Infants of Diabetic Mother
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Marina Abd Elsabour Adly, doctor, Assiut University
Other Study IDs: infants'congenital anomly
Record Dates: First submitted 2022-05-23; First posted 2022-05-26 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Congenital Abnormalities
MeSH Terms: conditions — Congenital Abnormalities

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional

INTERVENTIONS:
Device: Echo_CT_MRI_US_x ray — Examination: General and systemic examinations of the studied neonates. Investigation will be done to the neonates according to the clinical examination including imaging studies as X-rays, U/S, echocardiography, CT and MRI studies

SUMMARY:
The purpose of this study was to determine the pattern of congenital anomalies associated with maternal diabetes mellitus in newborns attending Assiut University children's Hospital.

DETAILED DESCRIPTION:
Infants of diabetic mothers have been shown in several studies to have an increased frequency of malformations. In previous studies, an increased frequency of several specific malformations has been noted, including anencephaly, bilateral renal agenesis, and double outlet right ventricle. Surveillance, used to identify all malformed infants in a consecutive sample of births, can identify a distinctive pattern of malformations among the affected infants.(1) Maternal pregestational diabetes mellitus is associated with an increased risk for congenital malformations of about2-4 times the background risk.(2) Perinatal outcome of the infant of the diabetic mother (IDM) depends on the onset, duration, and severity of maternal diabetes and is worse for IDM born from mothers with pre-existent insulin-dependent diabetes.(3) that glycemic control is associated with a reduced risk of congenital anomalies. However, the recommended threshold of HgA1c for pregestational diabetic women planning pregnancy is still not known.(4) Congenital anomalies are broadly classified into either single-system or multiple-system malformations. The first type affects a single organ system or body part,(5,6,7) and the second affects more than one organ system or body part. Major congenital anomalies are defined as those that, if uncorrected, could result in considerable impairment of the normal body functions or even reducing the life expectancy. Minor congenital anomalies include the anomalies that cause no disability or have no significant physical or functional effects and can be regarded as normal variants.(5,8,9) In another study conducted in Egypt on live-born babies, the incidence of minor congenital anomalies among infants of diabetic mothers was 18%, while the incidence was 11% for the major congenital anomalies, the later was 4.6 times higher than in the general population.(10) The pathophysiology of maternal diabetes induced birth defects is complex, however, clearly relates to maternal glucose levels. The mechanism is not entirely understood, but animal studies have shown it to be associated with decreased cell proliferation and increased cell apoptosis due to high oxidative stress, the second major change is altered gene expression causing deviation from the normal developmental process.(11) However, most congenital defects associated with diabetes occur in the cardiovascular, central nervous and musculoskeletal systems. Although hyperglycemia is a common mechanism for teratogenicity, differences in disease characteristics, such as age of onset, ethnicity, obesity and duration of disease, may affect the disease impact on the perinatal outcome and the rate of congenital anomalies.(11,12)

ELIGIBILITY:
Inclusion Criteria:

* The study will include all births of diabetic mothers

Exclusion Criteria:

* Other risk factors of congenital anomalies, such as TORCH infections, teratogenic drugs or irradiation.

Ages: 24 Days to 1 Year | Sex: All
Age Groups: Child
Study Population: The study will include all births of diabetic mothers
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2023-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
to determine the pattern of congenital anomalies associated with maternal diabetes mellitus in newborns | baseline
  Careful evaluation and early diagnosis of congenital anomalies in this high-risk group.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nasri HZ, Houde Ng K, Westgate MN, Hunt AT, Holmes LB. Malformations among infants of mothers with insulin-dependent diabetes: Is there a recognizable pattern of abnormalities? Birth Defects Res. 2018 Jan;110(2):108-113. doi: 10.1002/bdr2.1155. PMID 29377640
- [Background] Orbain MM, Johnson J, Nance A, Romeo AN, Silver MA, Martinez L, Leen-Mitchell M, Carey JC. Maternal diabetes-related malformations in Utah: A population study of birth prevalence 2001-2016. Birth Defects Res. 2021 Jan 15;113(2):152-160. doi: 10.1002/bdr2.1843. Epub 2020 Nov 23. PMID 33226174
- [Background] Ognean L, Boanta O, Visa G, Grosu F, Sofariu C, Gafencu M, Matei C, Iurian S. HYDROCEPHALY, SCHIZENCEPHALY, SPONDYLOCOSTAL DYSPLASIA, AND HYPOPARATHYROIDISM IN AN INFANT OF A DIABETIC MOTHER. Acta Endocrinol (Buchar). 2017 Oct-Dec;13(4):494-501. doi: 10.4183/aeb.2017.494. PMID 31149221
- [Background] Gabbay-Benziv R, Reece EA, Wang F, Yang P. Birth defects in pregestational diabetes: Defect range, glycemic threshold and pathogenesis. World J Diabetes. 2015 Apr 15;6(3):481-8. doi: 10.4239/wjd.v6.i3.481. PMID 25897357
- [Background] al-Gazali LI, Dawodu AH, Sabarinathan K, Varghese M. The profile of major congenital abnormalities in the United Arab Emirates (UAE) population. J Med Genet. 1995 Jan;32(1):7-13. doi: 10.1136/jmg.32.1.7. PMID 7897633
- [Background] Sawardekar KP. Profile of major congenital malformations at Nizwa Hospital, Oman: 10-year review. J Paediatr Child Health. 2005 Jul;41(7):323-30. doi: 10.1111/j.1440-1754.2005.00625.x. PMID 16014135
- [Background] Walden RV, Taylor SC, Hansen NI, Poole WK, Stoll BJ, Abuelo D, Vohr BR; National Institute of Child Health and Human Development Neonatal Research Network. Major congenital anomalies place extremely low birth weight infants at higher risk for poor growth and developmental outcomes. Pediatrics. 2007 Dec;120(6):e1512-9. doi: 10.1542/peds.2007-0354. Epub 2007 Nov 5. PMID 17984212
- [Background] Anyanwu LJC, Danborno B, Hamman WO. Birth prevalence of overt congenital anomalies in Kano Metropolis: overt congenital anomalies in the Kano. Uni J Pub Health. 2015;3(2):89-96.
- [Background] Kingston HM. ABC of clinical genetics. 3rd ed. London: BMJ Books; 2002.
- [Background] Ameen SK, Alalaf SK, Shabila NP. Pattern of congenital anomalies at birth and their correlations with maternal characteristics in the maternity teaching hospital, Erbil city, Iraq. BMC Pregnancy Childbirth. 2018 Dec 18;18(1):501. doi: 10.1186/s12884-018-2141-2. PMID 30563491
- [Background] Aberg A, Westbom L, Kallen B. Congenital malformations among infants whose mothers had gestational diabetes or preexisting diabetes. Early Hum Dev. 2001 Mar;61(2):85-95. doi: 10.1016/s0378-3782(00)00125-0. PMID 11223271
- [Background] Yang J, Cummings EA, O'connell C, Jangaard K. Fetal and neonatal outcomes of diabetic pregnancies. Obstet Gynecol. 2006 Sep;108(3 Pt 1):644-50. doi: 10.1097/01.AOG.0000231688.08263.47. PMID 16946226